CLINICAL TRIAL: NCT05847998
Title: Second Generation DICART Prototype Validation for Patients With Acute Circulatory Failure
Brief Title: Second Generation DICART Prototype Validation
Acronym: DICART II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL21_0635; 2021-A02595-36 (Other: IDRCB)
Record Dates: First submitted 2023-02-16; First posted 2023-05-08 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2024-03

CONDITIONS: Acute Circulatory Failure; Shock
Keywords: Acute Circulatory Failure; Shock; capillary refill time (CRT); prognosis; diagnostic; evaluation
MeSH Terms: conditions — Shock; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- measurement of capillary refill time (Experimental): measurement in a cohort of ICU adult patients with acute circulatory failure
  Interventions: Device: Standardized measurement of capillary refill time by second generation DICART prototype; Diagnostic Test: Clinical measurement of capillary refill time

INTERVENTIONS:
Device: Standardized measurement of capillary refill time by second generation DICART prototype — Capillary refill time is measured by two independent operators, each one blinded from the other, with second generation DICART prototype.
  Each operator performs two series of three consecutive measurement on the finger.
  Then, an operator performs a train of three measurements on the knee, and the other operator on the thorax
Diagnostic Test: Clinical measurement of capillary refill time — Capillary refill time is clinically measured by two independent operators, each one blinded from the other.
  Each operator performs, two series of three consecutive measurement on the second finger.
  Then, an operator performs a train of three measurements on the knee, and the other operator on the thorax, inverted relative to DICART measurements.

SUMMARY:
Capillary refill time (CRT) is a clinical sign for diagnosis of acute circulatory failure and response to treatment but is also associated with prognosis in patient with shock.

CRT is clinically evaluated by physician with a high risk of inter and intra evaluator variations, depending, for example, on measurement site, pressure applicated or visual evaluation.

The investigator hypothesizes that CRT measurement with second generation DICART prototype will be well correlated with clinical measurement.

ELIGIBILITY:
Inclusion Criteria:

->18 years old

* Acute circulatory failure
* Written informed consent given by patient or its relatives

Exclusion Criteria:

* Pregnant women, breastfeeding women, childbearing age women without oral contraception
* Cutaneous lesion at measurement site
* Patient under legal protection
* Patient already included in another interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-04-06 (Actual); Primary Completion 2023-10-28 (Actual); Study Completion 2023-10-28 (Actual)

PRIMARY OUTCOMES:
clinical capillary refill time measurement. | during procedure
  Intraclass correlation coefficient between clinical and automatic DICART capillary refill time measurement.
automatic DICART capillary refill time measurement. | during procedure
  Intraclass correlation coefficient between clinical and automatic DICART capillary refill time measurement.

SECONDARY OUTCOMES:
ROC curve with DICART device | during procedure
  ROC curve for DICART performance to detect a tissular hypoperfusion, defined as a clinical CRT superior to 3s
Inter-operator reproducibility in CRT measurement with DICART device | during procedure
  reproducibility in CRT measurement with DICART device using Bland-Altman comparison analysis
Inter-operator reproducibility in CRT measurement with clinical method | during procedure
  reproducibility in CRT measurement with DICART device using Bland-Altman comparison analysis
Intra-operator reproducibility in CRT measurement with DICART device | during procedure
  reproducibility in CRT measurement with DICART device using Bland-Altman comparison analysis
Intra-operator reproducibility in CRT measurement with clinical method | during procedure
  reproducibility in CRT measurement with DICART device using Bland-Altman comparison analysis
vital status | 30 days
  Association between CRT and 30 day survival without renal replacement therapy
survival rate without renal replacement therapy | 30 days
skin lesion assessed by clinical examination | during procedure
  Safety consideration about DICART use: qualitative skin examination
rash assessed by clinical examination | during procedure
  Safety consideration about DICART use: qualitative skin examination pain evaluation by numerical rating scale (0 means none and 3 severe)
pain evaluation by numerical rating scale | during procedure
  Safety consideration about DICART use: pain evaluation by numerical rating scale 0 corresponds to "no pain" and 10 to "worst pain imaginable".

CONTACTS AND LOCATIONS:
Overall Officials: Matthias JACQUET-LAGREZE, MD, PHD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Louis Pradel Cardiologic Hospistal, Bron, France

REFERENCES:
- [Result] Descamps A, Jacquet-Lagreze M, Aussal T, Fellahi JL, Ruste M. DiCARTTM device to measure capillary refill time: a validation study in patients with acute circulatory failure. J Clin Monit Comput. 2025 Oct;39(5):831-840. doi: 10.1007/s10877-025-01271-5. Epub 2025 Feb 26. PMID 40011397